CLINICAL TRIAL: NCT05500118
Title: Establishment of a Decision Aid Tool for Asymptomatic Small Leiomyoma and Analysis of Influencing Factors for Clinical Decision-making Using HIFU
Status: Recruiting | Type: Observational
Sponsor: Shenzhen Maternity & Child Healthcare Hospital (Other)
Responsible Party: Principal Investigator, Yu Dai, Associate Professor, Shenzhen Maternity & Child Healthcare Hospital
Other Study IDs: 2021KFKT030
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Leiomyoma, Uterine; High-Intensity Focused Ultrasound Ablation; Patients Decision Aids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- communication without PADs: We use traditional communication ways to discuss the conditions with patients.
- communication with PADs: The committee, composed of designers, doctors, nurses and patients, bases on guidelines and evidence-based medicine to make a tool. And we use this tool to discuss the conditions with patients.
  Interventions: Other: Patients Decision Aids

INTERVENTIONS:
Other: Patients Decision Aids — Patient Decision Aids (PDAs) are an important way to facilitate making decision by patients, helping patients make specific and prudent choices by providing information about treatment options and corresponding outcomes, including benefits and risks, related to their health status. The purpose of PDAs is to encourage patients to participate in decision-making. It makes it easier for patients and doctors to discuss treatment options. It effectively promotes communication between patients and doctors. It can help patients combine their own needs and professional advice to make better, more individualized diagnosis and treatment options.
  Groups: communication with PADs

SUMMARY:
With the younger patients diagnosed with asymptomatic leiomyoma, delay in the reproductive age of women, the advancement of medical technology, and the rapid development of treatment methods, there are many choices between gynecologists, gynecologists and patients because of experience and knowledge. It is not easy to make the most favorable choice for patients. This study is mainly led by a committee composed of designers, doctors, nurses and patients, and based on clinical guidelines and evidence-based medicine. Co-operating with patients with asymptomatic small leiomyoma, we want to find the influencing factors of clinical decision-making, and to establish a patient decision aid tool. We use prospective trial to verify that the use of this tool can improve patients' decision-making efficacy and further improve patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of leiomyoma: patients with leiomyoma diagnosed by imaging examinations (ultrasound and MRI) have no clinical symptoms;
2. Female with age in 18-55 years old;
3. The maximum diameter of a single leiomyoma is less than 5m, and the number does not exceed 10 by MRI;
4. No contraindications for sedation and analgesia;
5. Patients and their families agree to join this study, and can follow up on time.

Exclusion Criteria:

1. History of myomectomy, including transabdominal, laparoscopic, hysteroscopy, etc.;
2. History of connective tissue diseases or radiotherapy, especially abdominal radiotherapy;
3. With pregnancy, acute inflammation of the reproductive tract, or other gynecological benign and malignant diseases such as endometriosis and ovarian tumors;
4. The maximum diameter of leiomyoma is greater than or equal to 5cm;
5. Suspected malignant tumor, such as sarcoma;
6. Those with language communication barriers and unable to cooperate with sedative and analgesic programs;
7. Abdominal scarring, when diagnosed by ultrasound transabdominal scan, has obvious sound attenuation (more than 10mm range).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 18-55 years old woman diagnosed with uterine fibroids and without clinical symptoms
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-08-31 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction after using PDAs | 6-12 months
  The patients in PDAs will undertake the treatment by PDAs. And we will collect the satisfaction after 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Maternal and Child Health Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No